CLINICAL TRIAL: NCT00620542
Title: Study of Coronary Atheroma by Intravascular Ultrasound: Effect of Rosuvastatin Versus Atorvastatin (SATURN)
Brief Title: CRESTOR Athero Imaging Head to Head IVUS Study
Acronym: SATURN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D356IC00001; 2007-004000-13
Record Dates: First submitted 2008-02-06; First posted 2008-02-21 (Estimated); Results first posted 2012-06-25 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Atherosclerosis
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Rosuvastatin 20 mg (Experimental): Rosuvastatin 20 mg distributed in 2-week run-in period
  Interventions: Drug: Rosuvastatin
- Atorvastatin 40 mg (Active Comparator): Atorvastatin 40 mg distributed in 2-week run-in period
  Interventions: Drug: Atorvastatin
- Rosuvastatin 40 mg (Experimental): Rosuvastatin 40 mg distributed in core 2-year study
  Interventions: Drug: Rosuvastatin
- Atorvastatin 80 mg (Active Comparator): Atorvastatin 80 mg distributed in core 2-year study
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Rosuvastatin — capsule, oral, once daily
  Other Names: Crestor
  Arms: Rosuvastatin 20 mg; Rosuvastatin 40 mg
Drug: Atorvastatin — capsule, oral, one daily
  Other Names: Lipitor
  Arms: Atorvastatin 40 mg; Atorvastatin 80 mg

SUMMARY:
A 104-week, randomized, double-blind, parallel group, multi-center Phase IIIb study comparing the effects of treatment with rosuvastatin 40 mg or atorvastatin 80 mg on atherosclerotic disease burden as measured by intravascular ultrasound in patients with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indication for coronary angiography
* Angiographic evidence of Coronary Artery Disease (CAD), as defined by at least 1 lesion in a native coronary artery that has >20% reduction in lumen diameter by visual estimation
* Left main coronary artery must have <=50% reduction in lumen diameter by visual estimation
* LDL-C >100 mg/dL (2.6 mmol/L) for patients with no statin therapy in the past 4 weeks; LDL-C >80mg/dL (2.08mmol/L) for patients on therapy in the past 4 weeks

Exclusion Criteria:

* Use of certain lipid-lowering medication for more than 3 months within the previous 12 months. Longer periods of treatment are not permitted because of the potential effects of such therapy on coronary atherosclerosis.
* Patients who have symptoms consistent with moderate or greater severity of Congestive Heart Failure (CHF).
* Clinically significant heart disease which, in the opinion of the Principal Investigator (or designee), is likely to require coronary bypass surgery, cardiac transplantation, surgical repair and/or replacement during the course of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2333 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Nicholls, MBBS, PhD, Principal Investigator — Cleveland Clinic Foundation, Cardiovascular Medicine
Locations (195):
- United States (97):
  - Research Site, Huntsville, Alabama
  - Research Site, Los Angeles, California
  - Research Site, Mountain View, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Santa Rosa, California
  - Research Site, Torrance, California
  - Research Site, Boulder, Colorado
  - Research Site, Greeley, Colorado
  - Research Site, Loveland, Colorado
  - Research Site, Farmington, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Clearwater, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Melbourne, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Haven, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Elkhart, Indiana
  - Research Site, Hammond, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Merrillville, Indiana
  - Research Site, Valparaiso, Indiana
  - Research Site, Davenport, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, West Des Moines, Iowa
  - Research Site, Ashland, Kentucky
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Covington, Louisiana
  - Research Site, Bethesda, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, Takoma Park, Maryland
  - Research Site, Bay City, Michigan
  - Research Site, Grand Blanc, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Midland, Michigan
  - Research Site, Muskegon, Michigan
  - Research Site, Petoskey, Michigan
  - Research Site, Saginaw, Michigan
  - Research Site, Southfield, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Minneapolis, Minnesota
  - Research Site, Rochester, Minnesota
  - Research Site, Saint Cloud, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, New Brunswick, New Jersey
  - Research Site, Ridgewood, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, Johnson City, New York
  - Research Site, New York, New York
  - Research Site, Roslyn, New York
  - Research Site, Williamsville, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Gastonia, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Elyria, Ohio
  - Research Site, Kettering, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Perrysburg, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Tulsa, Oklahoma
  - Research Site, Bend, Oregon
  - Research Site, Eugene, Oregon
  - Research Site, Hillsboro, Oregon
  - Research Site, Danville, Pennsylvania
  - Research Site, Doylestown, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Wormleysburg, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Germantown, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Oak Ridge, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Bellevue, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
- Argentina (6):
  - Research Site, Buenos Aires, Buenos Aires
  - Research Site, Cap. Fed., Buenos Aires
  - Research Site, Ciudad de Buenos Aires, Buenos Aires
  - Research Site, Corrientes, Corrientes Province
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Rosario, Santa Fe-argentina
- Australia (5):
  - Research Site, Liverpool, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Chermside, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Perth, Western Australia
- Belgium (6):
  - Research Site, Aalst, Belgium
  - Research Site, Bruges, Belgium
  - Research Site, Brussels, Belgium
  - Research Site, Charleroi, Belgium
  - Research Site, Genk, Belgium
  - Research Site, Leuven, Belgium
- Brazil (8):
  - Research Site, Cariacica, Espírito Santo
  - Research Site, Vitória, Espírito Santo
  - Research Site, Goiânia, Goiás
  - Research Site, Cuiabá, Mato Grosso
  - Research Site, Uberlândia, Minas Gerais
  - Research Site, Curitiba, Paraná
  - Research Site, Ribeirão Preto, São Paulo
  - Research Site, São Paulo, São Paulo
- Canada (17):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Victoria, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Saint John, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saskatoon, Saskatchewan
- France (9):
  - Research Site, Besançon
  - Research Site, Bron
  - Research Site, Créteil
  - Research Site, Le Plessis-Robinson
  - Research Site, Marseille
  - Research Site, Pessac
  - Research Site, Quincy-sous-Sénart
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Szged
- Italy (9):
  - Research Site, Arezzo, AR
  - Research Site, Sesto San Giovanni, Milano
  - Research Site, Milan, MI
  - Research Site, Rozzano, MI
  - Research Site, Parma, PR
  - Research Site, Siena, SI
  - Research Site, Udine, UD
  - Research Site, Novara
  - Research Site, Roma
- Mexico (7):
  - Research Site, Aguascalientes, Aguascalientes
  - Research Site, Guadalajara, Jalisco
  - Research Site, D.F, Mexico
  - Research Site, Puebla City, Puebla
  - Research Site, Querétaro City, Querétaro
  - Research Site, Monterrey
  - Research Site, Tijuana
- Netherlands (10):
  - Research Site, Alkmaar
  - Research Site, Amsterdam
  - Research Site, Breda
  - Research Site, Eindhoven
  - Research Site, Enschede
  - Research Site, Leeuwarden
  - Research Site, Nieuwegein
  - Research Site, Nijmegen
  - Research Site, Rotterdam
  - Research Site, Zwolle
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Katowice
  - Research Site, Kędzierzyn-Koźle
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Zabrze
- Russia (5):
  - Research Site, Krasnogorsk, Moscow Oblast
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
  - Research Site, Tyumen
- Spain (6):
  - Research Site, Málaga, Andalusia
  - Research Site, Badalona, Catalonia
  - Research Site, Barcelona, Catalonia
  - Research Site, Madrid, Madrid
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Alicante, Valencia

REFERENCES:
- [Derived] Puri R, Nissen SE, Shao M, Ballantyne CM, Barter PJ, Chapman MJ, Erbel R, Libby P, Raichlen JS, Uno K, Kataoka Y, Nicholls SJ. Sex-related differences of coronary atherosclerosis regression following maximally intensive statin therapy: insights from SATURN. JACC Cardiovasc Imaging. 2014 Oct;7(10):1013-22. doi: 10.1016/j.jcmg.2014.04.019. Epub 2014 Sep 17. PMID 25240453
- [Derived] Puri R, Libby P, Nissen SE, Wolski K, Ballantyne CM, Barter PJ, Chapman MJ, Erbel R, Raichlen JS, Uno K, Kataoka Y, Tuzcu EM, Nicholls SJ. Long-term effects of maximally intensive statin therapy on changes in coronary atheroma composition: insights from SATURN. Eur Heart J Cardiovasc Imaging. 2014 Apr;15(4):380-8. doi: 10.1093/ehjci/jet251. Epub 2014 Jan 20. PMID 24448227
- [Derived] Puri R, Nissen SE, Libby P, Shao M, Ballantyne CM, Barter PJ, Chapman MJ, Erbel R, Raichlen JS, Uno K, Kataoka Y, Nicholls SJ. C-reactive protein, but not low-density lipoprotein cholesterol levels, associate with coronary atheroma regression and cardiovascular events after maximally intensive statin therapy. Circulation. 2013 Nov 26;128(22):2395-403. doi: 10.1161/CIRCULATIONAHA.113.004243. Epub 2013 Sep 16. PMID 24043299
- [Derived] Nicholls SJ, Ballantyne CM, Barter PJ, Chapman MJ, Erbel RM, Libby P, Raichlen JS, Uno K, Borgman M, Wolski K, Nissen SE. Effect of two intensive statin regimens on progression of coronary disease. N Engl J Med. 2011 Dec 1;365(22):2078-87. doi: 10.1056/NEJMoa1110874. Epub 2011 Nov 15. PMID 22085316

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2333 Coronary Artery Disease (CAD) patients with clinical indication for coronary angiography were randomized to Part A, the 2-week run-in period. Of these, 1578 patients were treated and 1385 completed Part A. The 1385 patients completing Part A were then randomized to Part B the core study period of 104 weeks of treatment.
Pre-assignment Details: Angiography was performed to determine if patients were qualified to continue in the study based on protocol-specified angiographic criteria. Patients who satisfied all inclusion and exclusion criteria had an Intravascular Ultrasound (IVUS) performed within 2 weeks of the qualifying angiography.
Groups:
- Rosuvastatin 20 mg; Atorvastatin 40 mg: 2 week run-in period
- Rosuvastatin 40 mg; Atorvastatin 80 mg: 2 year core study
Period: Part A (Run-in - 2 Weeks)
Arm/Group | Rosuvastatin 20 mg | Atorvastatin 40 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Started | 1167 (Of 1167 randomized, N=783 received treatment.) | 1166 (Of 1166 randomized, N=795 received treatment.) | 0 | 0
Received Treatment | 783 | 795 | 0 | 0
Completed | 695 | 690 | 0 | 0
Not Completed | 472 | 476 | 0 | 0
Not completed — Adverse Event | 12 | 15 | 0 | 0
Not completed — Protocol Violation | 406 | 409 | 0 | 0
Not completed — Withdrawal by Subject | 43 | 40 | 0 | 0
Not completed — Lost to Follow-up | 7 | 6 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Safety reasons | 0 | 1 | 0 | 0
Not completed — IVUS not available | 4 | 4 | 0 | 0
Period: Part B (2 Year Core Study)
Arm/Group | Rosuvastatin 20 mg | Atorvastatin 40 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Started | 0 | 0 | 694 (Of 694 patients randomized, N=691 received treatment.) | 691 (Of 691 patients randomized, N=689 received treatment.)
Received Treatment | 0 | 0 | 691 | 689
Intent-to-treat Population | 0 | 0 | 520 (Patients who received treatment and had a baseline and end of study (Week 104) IVUS) | 519 (Patients who received treatment and had a baseline and end of study (Week 104) IVUS)
Completed | 0 | 0 | 546 | 547
Not Completed | 0 | 0 | 148 | 144
Not completed — Adverse Event | 0 | 0 | 46 | 49
Not completed — Protocol Violation | 0 | 0 | 3 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 55 | 54
Not completed — Lost to Follow-up | 0 | 0 | 20 | 9
Not completed — Protocol Violation | 0 | 0 | 13 | 16
Not completed — Safety reasons | 0 | 0 | 2 | 3
Not completed — Study specific discontinuation criteris | 0 | 0 | 6 | 6
Not completed — IVUS not available | 0 | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Rosuvastatin 40 mg; Atorvastatin 80 mg: 2 years
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg | Total
Number analyzed (Participants) | 520 | 519 | 1039
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 402 | 395 | 797
  >=65 years | 118 | 124 | 242
Age Continuous [Mean (Standard Deviation); unit: years]
  Age (yrs) at Week 0 | 57.4 (8.60) | 57.9 (8.50) | 57.6 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 141 | 133 | 274
  Male | 379 | 386 | 765

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Study (Week 104) in Percent Atheroma Volume (PAV)
Description: Change in PAV computed as PAV(Week 104)-PAV(baseline) where PAV is calculated as:
  [sum(EEMcsa-LUMENcsa)/sum EEMcsa]*100 where EEMcsa is the cross-sectional area of the external elastic membrane and LUMENcsa is the cross-sectional area of the lumen, as measured by intravascular ultrasound IVUS of a coronary artery in patients with CAD.
Time Frame: End of study (Week 104)
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Median (95% Confidence Interval); unit: Percent change
Groups:
- Rosuvastatin 40 mg: Part B: Rosuvastatin 40 mg for core study - 2 years
- Atorvastatin 80 mg: Part B: Atorvastatin 80 mg for core study - 2 years
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 520 | 519
Percent change | -1.22 [-1.52 to -0.90] | -0.99 [-1.19 to -0.63]

2. Secondary Outcome: Numbers of Patients Showing Regression in PAV
Description: Regression defined as a change from baseline in PAV < 0
Time Frame: End of study (Week 104)
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 520 | 519
Participants | 356 | 328

3. Secondary Outcome: Change From Baseline to End of Study (Week 104) in Total Atheroma Volume (TAV)
Description: Change in TAV, as measured by IVUS, computed as TAV(Week 104)-TAV(baseline) where TAV is the sum(EEMcsa-LUMENcsa)/n. n is the number of cross-sections measured. TAV for each patient is calculated as the average area of atheroma per cross-section multiplied by the median number of cross-sections measured for all patients in the analysis population.
Time Frame: End of study (Week 104)
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Median (95% Confidence Interval); unit: mm^3
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 520 | 519
mm^3 | -6.39 [-7.52 to -5.12] | -4.42 [-5.98 to -3.26]

4. Secondary Outcome: Numbers of Patients Showing Regression in TAV
Description: Regression defined as a change from baseline in TAV < 0
Time Frame: End of study (Week 104)
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Number; unit: Participants
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 520 | 519
Participants | 371 | 336

5. Secondary Outcome: Total Cholesterol Blood Level
Description: Time-weighted average is calculated as the lipid value times the number of days since last lipid assessment, summed for all and divided by the number of days from Part B randomization to date of the last lipid evaluation.
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 519 | 519
mg/dL | 139.38 (1.24) | 144.05 (1.23)

6. Secondary Outcome: LDL-C Blood Level
Description: as for outcome 5
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 519 | 519
mg/dL | 62.64 (1.00) [lower limit 1.00] | 70.18 (0.99) [lower limit 0.99]

7. Secondary Outcome: HDL-C Blood Level
Description: as for outcome 5
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 519 | 519
mg/dL | 50.43 (0.54) [lower limit 0.54] | 48.64 (0.53) [lower limit 0.53]

8. Secondary Outcome: Triglycerides Blood Level
Description: as for outcome 5
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 519 | 519
mg/dL | 132.50 (2.44) [lower limit 2.44] | 126.58 (2.43) [lower limit 2.43]

9. Secondary Outcome: Non-HDL-C Blood Level
Description: as for outcome 5
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 519 | 519
mg/dL | 88.95 (1.15) [lower limit 1.15] | 95.41 (1.14) [lower limit 1.14]

10. Secondary Outcome: LDL-C/HDL-C Blood Level
Description: as for outcome 5
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 519 | 519
Ratio | 1.30 (0.02) [lower limit 0.02] | 1.50 (0.02) [lower limit 0.02]

11. Secondary Outcome: Total Cholesterol/HDL-C Blood Level
Description: as for outcome 5
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 519 | 519
Ratio | 2.88 (0.03) [lower limit 0.03] | 3.08 (0.03) [lower limit 0.03]

12. Secondary Outcome: Non-HDL-C/HDL-C Blood Level
Description: as for outcome 5
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 519 | 519
Ratio | 1.88 (0.03) [lower limit 0.03] | 2.08 (0.03) [lower limit 0.03]

13. Secondary Outcome: Apolipoprotein B Blood Level
Description: as for outcome 5
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 518 | 519
mg/dL | 72.55 (0.85) [lower limit 0.85] | 75.12 (0.85) [lower limit 0.85]

14. Secondary Outcome: Apolipoprotein A-1 Blood Level
Description: as for outcome 5
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 518 | 519
mg/dL | 146.81 (1.03) [lower limit 1.03] | 137.68 (1.02) [lower limit 1.02]

15. Secondary Outcome: Apoliprotein B/Apolipoprotein A-1 Blood Level
Description: as for outcome 5
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: Ratio
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 518 | 519
Ratio | 0.51 (0.01) | 0.56 (0.01)

16. Secondary Outcome: VLDL-C During the 104 Week Treatment Period
Description: as for outcome 5
Time Frame: 104 weeks
Population: Intent-to-Treat population (patients received at least one dose of study drug and had pre-study and post-study IVUS).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Rosuvastatin 40 mg | Atorvastatin 80 mg
Number analyzed (Participants) | 519 | 519
mg/dL | 26.05 (0.45) | 25.03 (0.44)

ADVERSE EVENTS:
Arm/Group | Rosuvastatin 20 mg | Atorvastatin 40 mg | Rosuvastatin 40 mg | Atorvastatin 80 mg
Serious Adverse Events (participants affected / at risk) | 21/783 | 25/795 | 194/691 | 168/689
Other Adverse Events (participants affected / at risk) | 0/783 | 0/795 | 210/691 | 213/689
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 20 mg (N=783) | Atorvastatin 40 mg (N=795) | Rosuvastatin 40 mg (N=691) | Atorvastatin 80 mg (N=689)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 5 | 5 | 25 | 28
Angina Unstable (Cardiac disorders) | 0 | 2 | 17 | 11
Coronary Artery Stenosis (Cardiac disorders) | 1 | 0 | 12 | 9
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 10 | 4
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1 | 5 | 6
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 3 | 6
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 5 | 3
Mitral Valve Incompetence (Cardiac disorders) | 0 | 0 | 3 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 3
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0 | 2 | 2
Bradycardia (Cardiac disorders) | 0 | 2 | 1 | 2
Myocardial Ischaemia (Cardiac disorders) | 0 | 0 | 2 | 0
Sick Sinus Syndrome (Cardiac disorders) | 0 | 0 | 1 | 2
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 0 | 1 | 1
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary Artery Insufficiency (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary Artery Thrombosis (Cardiac disorders) | 0 | 0 | 1 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial Rub (Cardiac disorders) | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 1 | 1
Sinus Arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 0 | 0 | 0 | 1
Congenital Coronary Artery Malformation (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Hip Dysplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Vertigo Positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Basedow's Disease (Endocrine disorders) | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Retinal Detachment (Eye disorders) | 0 | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Colonic Polyp (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Erosive Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric Polyps (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Retroperitoneal Haematoma (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 1 | 3 | 14 | 7
Chest Pain (General disorders) | 0 | 0 | 7 | 7
Chest Discomfort (General disorders) | 0 | 0 | 1 | 0
Device Malfunction (General disorders) | 0 | 0 | 1 | 0
Device Occlusion (General disorders) | 0 | 0 | 1 | 0
Device Stimulation Issue (General disorders) | 0 | 0 | 1 | 0
Hernia Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0
Sudden Death (General disorders) | 0 | 0 | 0 | 1
Thrombosis In Device (General disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 4 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 4 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 3 | 2
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 2 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 1
Appendicitis Perforated (Infections and infestations) | 0 | 0 | 1 | 0
Arthritis Bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Dengue Fever (Infections and infestations) | 0 | 0 | 1 | 0
Groin Infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes Zoster Infection Neurological (Infections and infestations) | 0 | 0 | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 1
Pilonidal Cyst (Infections and infestations) | 0 | 0 | 1 | 0
Puncture Site Infection (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 6 | 3
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Fractured Coccyx (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Heat Exhaustion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
In-Stent Arterial Restenosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post Procedural Myocardial Infarction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 0 | 2
Cardiac Stress Test Abnormal (Investigations) | 1 | 0 | 0 | 0
Heart Rate Irregular (Investigations) | 0 | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 0 | 0 | 0 | 1
Occult Blood Positive (Investigations) | 0 | 0 | 1 | 0
Transaminases Increased (Investigations) | 0 | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Bone Loss (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Floating Patella (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 2
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Colon Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Extranodal Marginal Zone B-Cell Lymphoma (Malt Type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Eyelid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Neoplasm Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Throat Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 3 | 6
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 3
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 2 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 2 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 2
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 2 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 2 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Complicated Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Grand Mal Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhagic Stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Intracranial Hypotension (Nervous system disorders) | 0 | 0 | 0 | 1
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 0 | 1
Dependence (Psychiatric disorders) | 0 | 0 | 0 | 1
Panic Attack (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 3 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 2
Bladder Neck Obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Calculus Bladder (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureteric Stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal Obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 0 | 0 | 1 | 0
Intermittent Claudication (Vascular disorders) | 0 | 0 | 2 | 1
Subclavian Artery Stenosis (Vascular disorders) | 0 | 0 | 2 | 0
Aortic Stenosis (Vascular disorders) | 0 | 0 | 1 | 0
Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 0 | 1
Arterial Stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 1 | 0
Femoral Arterial Stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1
Iliac Artery Stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis Superficial (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin 20 mg (N=783) | Atorvastatin 40 mg (N=795) | Rosuvastatin 40 mg (N=691) | Atorvastatin 80 mg (N=689)
ANGINA PECTORIS (Cardiac disorders) | 0 | 0 | 61 | 65
FATIGUE (General disorders) | 0 | 0 | 32 | 39
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 99 | 91
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 50 | 43
HYPERTENSION (Vascular disorders) | 0 | 0 | 36 | 40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less